CLINICAL TRIAL: NCT05997992
Title: Clinical Efficacy Evaluation of Electroacupuncture as Adjuvant Therapy for Female Patients With Overactive Bladder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11-XD-071
Record Dates: First submitted 2023-01-29; First posted 2023-08-18 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Overactive Bladder
Keywords: Urge Incontinence; Overactive bladder; quality of life; TCM constitution,; Electroacupuncture
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — Electroacupuncture

STUDY DESIGN:
Intervention Model Description: The research is a single-blind randomized controlled human trial.The research is a single-blind randomized controlled human trial. It is planned to select 100 women aged 20-80 years with a diagnosis of OAB in outpatient clinics, and divide them into an experimental group and a control group of 50 each. The experimental group received electroacupuncture at Baihui(GV20), bilateral Sanyinjiao(SP-6) and Fuliu points(KP-7); the control group received placebo acupuncture
Who Masked: Participant
Masking Description: The research is a single-blind randomized controlled human trial.The participant will divide into control group or experimental group randomly by random number table.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Electroacupuncture group (Experimental): The Electroacupuncture group received electroacupuncture at Baihui(GV20), bilateral Sanyinjiao(SP-6) and Fuliu points(KP-7).20 minutes of acupuncture.
  Twice a week.
  Interventions: Device: electroacupuncture
- Sham acupuncture group (Placebo Comparator): The control group received placebo acupuncture.Except for placebo acupuncture, which won't penetrate the skin, the rest is the same as the Electroacupuncture group.
  Interventions: Device: sham acupuncture

INTERVENTIONS:
Device: electroacupuncture — Electroacupuncture is a form of acupuncture where a small electric current is passed between pairs of acupuncture needles. According to some acupuncturists, this practice augments the use of regular acupuncture, can restore health and well-being, and is particularly good for treating pain.
  Arms: Electroacupuncture group
Device: sham acupuncture — Acupuncture does not penetrate the skin, and the electroacupuncture machine is not plugged in.
  Arms: Sham acupuncture group

SUMMARY:
Overactive bladder (OAB) is often accompanied by frequent urination and nocturia, and does not necessarily manifest as urge incontinence. Urgency to urinate and frequent urination can lead to psychological burdens, affect interpersonal relationships and reduce women's quality of life.

Treatment of OAB includes lifestyle changes, behavioral therapy, drug therapy, neuromodulation, botulinum toxin therapy, and surgical intervention. At present, anticholinergic drugs are usually the first-line treatment for OAB, but the side effects of dry mouth often lead to poor patient compliance.

Transcutaneous tibial nerve stimulation (PTNS) is a minimally invasive neuromodulation technique. Past studies have confirmed that PTNS has clinical efficacy in treating symptoms related to overactive bladder, while TCM's electroacupuncture is similar to PTNS. The main purpose of this study was to evaluate the specific acupoints in accordance with traditional Chinese medicine theory in women with OAB under conventional Western medicine treatment to evaluate the improvement of women's related urinary tract symptoms, quality of life and autonomic nervous system function.

DETAILED DESCRIPTION:
Overactive bladder (OAB) is often accompanied by frequent urination and nocturia, and does not necessarily manifest as urge incontinence. Urgency to urinate and frequent urination can lead to psychological burdens, affect interpersonal relationships and reduce women's quality of life.

Treatment of OAB includes lifestyle changes, behavioral therapy, drug therapy, neuromodulation, botulinum toxin therapy, and surgical intervention. At present, anticholinergic drugs are usually the first-line treatment for OAB, but the side effects of dry mouth often lead to poor patient compliance.

Transcutaneous tibial nerve stimulation (PTNS) is a minimally invasive neuromodulation technique. Past studies have confirmed that PTNS has clinical efficacy in treating symptoms related to overactive bladder, while TCM's electroacupuncture is similar to PTNS. The main purpose of this study was to evaluate the specific acupoints in accordance with traditional Chinese medicine theory in women with OAB under conventional Western medicine treatment to evaluate the improvement of women's related urinary tract symptoms, quality of life and autonomic nervous system function.

ELIGIBILITY:
Inclusion Criteria:

* Female patient aged 20-80 with overactive bladder.

Exclusion Criteria:

* Patient has history of cancer, stroke, or hyperthyroidism..
* Patient isn't willing to accept acupuncture or moxibustion treatment.
* Patient who is pregnant or plan to pregnant.
* Patient with urinary tract infection.
* Patient who had injection of botulinum toxin (Botox®), PTNS or SMN treatment before.
* Patient recieved acupuncture treatment before.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Urinary tract related questionnair | Study spans 8 weeks: initial data collection, biweekly collections, 1-week break after 6 weeks, final collection in week 8. 5 questionnaire rounds in total. Proposed timeline.
  Measuring OAB scores to record the differ between two groups and time.Higher scores indicate more severe symptoms of overactive bladder syndrome.
King's Health Quality of Life Questionnaire(KHQ) | Study spans 8 weeks: initial data collection, biweekly collections, 1-week break after 6 weeks, final collection in week 8. 5 questionnaire rounds in total. Proposed timeline.
  Measuring KHQ scores to record the differ between two groups and time.Higher scores indicate more significant impact of bladder-related issues on quality of life.
Heart rate variability(HRV) | Study spans 8 weeks: initial data collection, biweekly collections, 1-week break after 6 weeks, final collection in week 8. 5 questionnaire rounds in total. Proposed timeline.
  Measuring HRV to record the differ between two groups and time.Whether the balance of the autonomic nervous system in HRV can also be used to infer the severity of OAB symptoms is also an observation target for the researchers.

SECONDARY OUTCOMES:
Is the dose of the drug reduced? | Every week will record the dose that participants take.A total of 8 weeks.
  We record the doses of drugs that participants take.By comparing the differences in medication dosage over the course of 8 weeks, we aim to investigate the effectiveness of the therapeutic intervention.
Are the side effects reduced? | Every week will record side effects of taking medicine.A total of 8 weeks.
  We record participants' side effects after taking the drug.By comparing the differences in side effects over the course of 8 weeks, we aim to explore the effectiveness of the therapeutic intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Buddhist Taipei Tzu Chi General Hospital, New Taipei City, Taiwan